CLINICAL TRIAL: NCT06543875
Title: Overweight, Obesity and Weight Variation Among Incarcerated Women in French Guiana: a Study of Factors Associated With Weight Gain
Acronym: PPFCPG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: PPFCPG
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women incarcerated at the Penitentiary Center of French Guiana

SUMMARY:
Overweight and obesity are a public health issue, given the morbi-mortality they entail: increase in chronic diseases such as cardiovascular disease, diabetes, musculoskeletal disorders, certain cancers.

According to the 2019 European Health Survey, French Guiana has a high rate of overweight and obesity, affecting 51% of its population (compared with 47% in mainland France), with a higher prevalence among women (23%), this phenomenon being partly attributed to unfavorable eating habits and a sedentary lifestyle. Another study in French Guiana showed that 54.7% of those surveyed were overweight or obese, with a higher risk of obesity among single women, often from non-French Caribbean and South American immigrant backgrounds, unemployed or poorly educated. Some of these risk factors are found in the general prison population: immigrant population, unemployed, low socio-educational level.

A meta-analysis published in 2017 analyzed weight variations in individuals during their period of incarceration. All but one study reported an increase in BMI and weight gain, in a significant proportion of participants. Weight gain was associated with gender, and was higher in women. A systematic review of 2020 on cardiovascular risks associated with incarceration revealed, through meta-regression, a mean weight increase of 5.3 kg (CI95%: 0.5 to 10.1) and a variation in Body Mass Index (BMI) of 1.8 kg/m2 (CI95%: -0.9 to 4.6) after two years of incarceration, attributed to a sedentary lifestyle, inappropriate diet, forced smoking cessation, use of psychotropic medication and high levels of stress.

The higher prevalence of obesity among women is a trend observed both in French Guiana and in the prison environment, where weight gain is associated with the female gender. There are currently no studies examining the weight of female prisoners in French Guiana, its evolution and the identification of risk factors linked to weight gain in the CPG.

ELIGIBILITY:
Inclusion Criteria:

Female adult in prison for more than 7 days at the time of the interviews

Exclusion Criteria:

* Refusal to participate
* Cognitive impairment or lack of communication resulting in inability to complete questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Exhaustive selection method including all women incarcerated at the prison when the interviews were conducted.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
overall weight of women incarcerated | from date of incarceration until the date of inclusion, at least 7 days and no upper limit
  This variation is calculated by subtracting the initial weight on entry into the current weight at the time of the interview. T Weight measurements are taken in kilograms (kg to one decimal place) at two decimal place) at two key points: o These measurements are valid and reproducible: weight taken on a standardized scale scale, in light clothing and barefoot,
  The primary endpoint will quantify changes in weight I during the period of incarceration, and will serve as a basis for to assess the impact of various factors on weight gain in female women prisoners.
overall BMI trends of women incarcerated | from date of incarceration until the date of inclusion, at least 7 days and no upper limit
  This variation is calculated by subtracting the initial weight on entry into the current weight at the time of the interview for BMI.
  Weight measurements are taken in kilograms (kg to one decimal place) at two decimal place) at two key points: on entry into detention and at the time of the and during the interview, based on medical records and individual individual interviews.
  BMI will be calculated using weight and height: calculation of body mass index (BMI) body mass index (BMI): weight (kg) / height (m2).

SECONDARY OUTCOMES:
1) Study changes in weight over time | from date of incarceration until the date of inclusion, at least 7 days and no upper limit
  Intermediate weights (kg to one decimal place) available in the medical record between entry into detention and inclusion will be recorded This will enable a more precise study of changes in weight as a function of time and length of incarceration. The frequency with which intermediate weights are recorded in a woman's medical record may vary from one patient, as they are not systematically recorded during medical consultations, when they take place.
1) Study changes in BMI over time | from date of incarceration until the date of inclusion, at least 7 days and no upper limit
  Intermediate weights (kg to one decimal place) available in the medical record between entry into detention and inclusion will be recorded, and intermediate BMIs calculated. This will enable a more precise study of changes in weight and BMI as a function of time and length of incarceration. The frequency with which intermediate weights are recorded in a woman's medical record may vary from one patient, as they are not systematically recorded during medical consultations, when they take place.
prevalence of overweight and obesity, including those at high risk of metabolic and vascular disease: | from date of incarceration until the date of inclusion, at least 7 days and no upper limit
  On the one hand, at entry into detention, and on the other, at inclusion. Calculation of body mass index (BMI): weight (kg) / height (m2).
  Interpretation of BMI according to WHO recommendations:
  * < 18.5 kg/m²: underweight ;
  * = or > 18.5 and < 25 kg/m²: normal build;
  * = or > 25 and < 30 kg/m²: overweight;
  * = or > 30 kg/m²: obese; Waist circumference will be measured in cm during the interview only, using a tape measure (midway between the lower edge of the last palpable rib and the top of the iliac crest, with a tape measure placed horizontally, at the end of a normal exhalation according to the Belgian Association for the Study of Obesity recommended by HAS). HAS classification: high waist circumference in women when >/= 80 cm.
3) Describe the population of female inmates incarcerated | from date of incarceration until the date of inclusion, at least 7 days and no upper limit
  collect socio-demographic and economic data, lifestyle habits, medical history, medication intake, using the medical record and questionnaire. Judicial information :
  Socio-demographic information :
  Clinical information :
  Habitus information :
  Medical information :
factors associated with weight gain during incarceration: Comparison between women who have gained weight, to those who have not gained weight | from date of incarceration until the date of inclusion, at least 7 days and no upper limit
  Weight gain is evidenced by by an increase in BMI >/= 1 point (or definition of a delta in of a delta in kilograms).
  a Questionnaire will be carried out during the interview with the patient. Results concerning the following variable will be aggregated in order to identify which factor is implicated in weight change between physical activity, sleep quantity and quality, eating habits, habits linked to incarceration, number of female cellmates cell, presence of intra- and extra-custodial contacts access to visiting room and telephone, whether or not trial has been completed, work at CPG

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, Guyane Française, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided